CLINICAL TRIAL: NCT05192733
Title: An International, Multisociety Practice Survey Of Extubation Following Elective Infratentorial Craniotomy In Adult Neurosurgical Patients
Brief Title: PRICE Survey Of Extubation Following Infratentorial Craniotomy
Acronym: PRICE1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Hervé Quintard (Unknown); Torstein Meling (Unknown); Nicolai Goettel (Unknown); Lien Jakus (Unknown); Camille Levy (Unknown)
Responsible Party: Principal Investigator, John Gaudet, Chef de Clinique en Anesthésie, Centre Hospitalier Universitaire Vaudois
Other Study IDs: Req-2021-01236
Record Dates: First submitted 2021-12-13; First posted 2022-01-14 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Infratentorial Neoplasms
Keywords: Airway Extubation; Prediction; Prevalence; Survey
MeSH Terms: conditions — Infratentorial Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Specialty: We will compare responses across the following clinical specialties :
  1. Neuroanesthesiologists
  2. Neurosurgeons
  3. Neurocritical care specialists NB: Some participants may have a double clinical specialty.
  Interventions: Other: Survey
- Clinical Setting: We will compare responses across the following clinical settings:
  1. Cities
  2. Countries
  3. Number of cases per year
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — This is a cross-sectional practice survey. There is no intervention.

SUMMARY:
The PRICE study primarily aims to identify predictors of early extubation following elective infratentorial craniotomy in adults. It also aims to (i) measure the rate of early extubation in different clinical settings; and (ii) study how the decision to extubate early is made and communicated in clinical practice. The first phase of the study (PRICE1) is a brief online survey addressed to physicians in charge of neurosurgical patients (neuroanesthesiologists, neurosurgeons, neurocritical care specialists) in multiple countries.

ELIGIBILITY:
Inclusion Criteria:

* Physician actively involved in delivering care to neurosurgical patients
* Physician formerly involved in delivering care to neurosurgical patients

Exclusion Criteria:

* Has already completed the survey

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physicians involved in delivering care to neurosurgical patients: neuroanesthesiologists, neurosurgeons, neurocritical care specialists
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of early extubation | 3 months
  Percentage of patients being extubated early, as estimated by responders. Early extubation is defined as extubation at the end of surgery, in the operating room, prior to discharge to recovery or intensive care.

SECONDARY OUTCOMES:
Inventory of perceived main predictors of early extubation | 3 months
  Participants to the survey can select up to 3 of the following options:
  Survey options are:
  Patient's level of consciousness Evidence of brainstem dysfunction Patient's physical status prior to surgery History or suspicion of difficult airway Preoperative imaging Duration of surgery Course of surgery Time of day when surgery ends Other (to be completed by responder)
Personnel perceived to make the decision to extubate early | 3 months
  Participants to the survey can select 1 or several of the following options:
  Anesthesiologist Neurosurgeon Neurocritical care physician

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Cata JP, Saager L, Kurz A, Avitsian R. Successful extubation in the operating room after infratentorial craniotomy: the Cleveland Clinic experience. J Neurosurg Anesthesiol. 2011 Jan;23(1):25-9. doi: 10.1097/ANA.0b013e3181eee548. PMID 21252705
- [Background] Cai YH, Wang HT, Zhou JX. Perioperative Predictors of Extubation Failure and the Effect on Clinical Outcome After Infratentorial Craniotomy. Med Sci Monit. 2016 Jul 12;22:2431-8. doi: 10.12659/msm.899780. PMID 27404044